CLINICAL TRIAL: NCT01190085
Title: Effects of Ghrelin on Alcohol Cue Reactivity and Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Lorenzo Leggio, Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 1005000183
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Alcoholism
Keywords: alcoholism; ghrelin; craving
MeSH Terms: conditions — Alcoholism | interventions — Ghrelin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ghrelin (1 microg/kg) (Active Comparator): A 1 microg/kg dose of intravenous human acetylated ghrelin was administered once approximately 10 minutes before the start of the alcohol cue-reactivity experiment.
  Interventions: Drug: Ghrelin
- Ghrelin (3 microg/kg) (Active Comparator): A 3 microg/kg dose of intravenous human acetylated ghrelin was administered once approximately 10 minutes before the start of the alcohol cue-reactivity experiment.
  Interventions: Drug: Ghrelin
- Saline Solution (Placebo Comparator): Intravenous saline solution (matched placebo) was administered once approximately 10 minutes before the start of the alcohol cue-reactivity experiment.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Ghrelin — A 1 microg/kg dose of intravenous human acetylated ghrelin was administered once approximately 10 minutes before the start of the alcohol cue-reactivity experiment.
  Other Names: human acetylated ghrelin
  Arms: Ghrelin (1 microg/kg)
Drug: Ghrelin — A 3 microg/kg dose of intravenous human acetylated ghrelin was administered once approximately 10 minutes before the start of the alcohol cue-reactivity experiment.
  Other Names: human acetylated ghrelin
  Arms: Ghrelin (3 microg/kg)
Drug: Saline solution — Intravenous saline solution (matched placebo) was administered once approximately 10 minutes before the start of the alcohol cue-reactivity experiment.
  Other Names: matched placebo
  Arms: Saline Solution

SUMMARY:
Only a few medications are approved for the treatment of alcohol dependence and there exists a substantial need for discovering ways to provide more effective treatments. Accordingly, identifying new potential neuropharmacological targets in the treatment of alcohol dependence represents a high priority in public health. Ghrelin is a 28-amino acid peptide acting as the endogenous ligand for the growth hormone secretagogue receptor (GHS-R). Ghrelin was first isolated from the stomach, but a central hypothalamic production of ghrelin has also been demonstrated. Ghrelin plays a key role in the regulation of appetite. Consistent with the common neurobiological substrates for control of food and alcohol consumption, preclinical investigations suggest that ghrelin plays a role in the neurobiology of alcohol dependence, thus representing a new potential neuropharmacology target. In keeping with the preclinical studies, human investigations showed that alcohol consumption affects blood ghrelin levels and that blood ghrelin levels significantly and positively correlate with craving measurements in alcohol-dependent individuals. The effects of exogenous ghrelin injected intravenous (i.v.) in alcohol-dependent individuals, however, have never been investigated. The current project proposes a randomized double-blind placebo-controlled 3-group between-subject laboratory study aimed at investigating the effects of exogenous ghrelin i.v. on non-treatment seeking alcohol-dependent subjects in terms of urges to drink, attention to cues and related psychophysiological measures. This project has the goals to: i) conduct an alcohol laboratory study testing the role of ghrelin i.v., therefore demonstrating the feasibility of such a study and the safety of ghrelin i.v. when administered to alcohol-dependent individuals; and ii) explore the effects of ghrelin i.v. on alcohol craving assessed under controlled conditions, such as a cue-reactivity (CR) experiment.

This study will address whether alcohol craving is affected when ghrelin levels are modified acutely via a ghrelin i.v. injection. Given the crucial need to expand our understanding of the underlying neurobiology of alcoholism, this study potentially will lead to identify new targets for the development of pharmacological treatments that may improve interventions for alcohol dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

* Understanding that this is not a treatment study.
* Breath alcohol concentration (BAC) equal to 0.00 when the participants sign the informed consent document.
* Age between 18 and 70 years old (inclusive).
* Female participants must be postmenopausal for at least one year, surgically sterile, or practicing an effective method of birth control before entry and throughout the study; have a negative urine pregnancy test at screening and cue-reactivity (CR) visits.
* Diagnosis of Alcohol dependence using Module E of the structured clinical interview for the Diagnostic and Statistical Manual of Mental Disorders - Text Revised (DSM-IV-TR).
* Participants must meet criteria for heavy drinking, defined as averaging ≥4 drinks/day for women and ≥5 drinks/day for men during a consecutive 30-day period within the 90 days prior to baseline evaluation
* Good health as confirmed by medical history, physical examination, electrocardiogram (ECG), laboratory tests and vital signs.
* Participant must be willing to receive an I.V. line.

Exclusion Criteria:

* Individuals expressing interest in treatment for alcoholism.
* Females who are of child bearing potential and not practicing effective birth control.
* Current (last 12 months) diagnosis of dependence on any psychoactive substance other than alcohol and nicotine (according to the DSM-IV-TR)
* DSM-IV-TR Axis I criteria for a lifetime diagnosis of schizophrenia, bipolar disorder, or other psychoses; an active illness within the past 6 months that meet the DSM-IV-TR criteria for a diagnosis of Major Depressive Disorder or Anxiety Disorder; in the investigators' opinion, moderate to severe risk of suicide (e.g. active plan, or attempt in last 6 months).
* History of hospitalization for alcohol intoxication delirium, alcohol withdrawal delirium or seizure.
* Clinical Institute Withdrawal Assessment for Alcohol revised (CIWA-Ar) ≥ 10, at any assessment.
* Positive urine drug screen at baseline for any illegal substance other than marijuana (a urine drug screen may be repeated once during the screening period).
* Subjects who have received any behavioral and/or pharmacological treatment for alcoholism within the past 30 days.
* Current use of psychotropic medications that cannot be discontinued.
* Clinically significant medical abnormalities [e.g., alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >300% the upper limit of normal].
* Significant medical conditions, such as cancer, liver cirrhosis, heart chronic failure, chronic kidney failure, chronic intestinal diseases (e.g., Crohn's disease), chronic neurological disorders (e.g., tardive dyskinesia, epilepsy, Parkinson's disease), diabetes, obesity [Body Mass Index(BMI) ≥ 30 kg/m2].
* Participants with a history of hypotension clinically significant (e.g.: history of fainting and/or syncopal attacks).
* No history of adverse reactions or hypersensitivity to ghrelin i.v. nor history of adverse reactions to needle puncture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

REFERENCES:
- [Background] Leggio L. Role of the ghrelin system in alcoholism: Acting on the growth hormone secretagogue receptor to treat alcohol-related diseases. Drug News Perspect. 2010 Apr;23(3):157-66. doi: 10.1358/dnp.2010.23.3.1429490. PMID 20440417
- [Background] Addolorato G, Capristo E, Leggio L, Ferrulli A, Abenavoli L, Malandrino N, Farnetti S, Domenicali M, D'Angelo C, Vonghia L, Mirijello A, Cardone S, Gasbarrini G. Relationship between ghrelin levels, alcohol craving, and nutritional status in current alcoholic patients. Alcohol Clin Exp Res. 2006 Nov;30(11):1933-7. doi: 10.1111/j.1530-0277.2006.00238.x. PMID 17067359
- [Background] Jerlhag E, Egecioglu E, Landgren S, Salome N, Heilig M, Moechars D, Datta R, Perrissoud D, Dickson SL, Engel JA. Requirement of central ghrelin signaling for alcohol reward. Proc Natl Acad Sci U S A. 2009 Jul 7;106(27):11318-23. doi: 10.1073/pnas.0812809106. Epub 2009 Jun 29. PMID 19564604
- [Background] Leggio L, Addolorato G, Cippitelli A, Jerlhag E, Kampov-Polevoy AB, Swift RM. Role of feeding-related pathways in alcohol dependence: A focus on sweet preference, NPY, and ghrelin. Alcohol Clin Exp Res. 2011 Feb;35(2):194-202. doi: 10.1111/j.1530-0277.2010.01334.x. Epub 2010 Nov 8. PMID 21058960
- [Background] Leggio L, Ferrulli A, Cardone S, Nesci A, Miceli A, Malandrino N, Capristo E, Canestrelli B, Monteleone P, Kenna GA, Swift RM, Addolorato G. Ghrelin system in alcohol-dependent subjects: role of plasma ghrelin levels in alcohol drinking and craving. Addict Biol. 2012 Mar;17(2):452-64. doi: 10.1111/j.1369-1600.2010.00308.x. Epub 2011 Mar 11. PMID 21392177
- [Result] Leggio L, Zywiak WH, Fricchione SR, Edwards SM, de la Monte SM, Swift RM, Kenna GA. Intravenous ghrelin administration increases alcohol craving in alcohol-dependent heavy drinkers: a preliminary investigation. Biol Psychiatry. 2014 Nov 1;76(9):734-41. doi: 10.1016/j.biopsych.2014.03.019. Epub 2014 Mar 25. PMID 24775991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited via advertisements in local public transportation and mass-media
Period: Overall Study
Arm/Group | Ghrelin (1 Microg/kg) | Ghrelin (3 Microg/kg) | Saline Solution
Started | 13 | 14 | 18
Completed | 13 | 14 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ghrelin (1 Microg/kg) | Ghrelin (3 Microg/kg) | Saline Solution | Total
Number analyzed (Participants) | 13 | 14 | 18 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 18 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (9.8) | 43.9 (8.6) | 46.6 (9.0) | 44.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 7 | 16
  Male | 9 | 9 | 11 | 29
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 18 | 45

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Visual Analogue Scale (A-VAS)
Description: Whether ghrelin intravenous (i.v.), as compared to saline i.v., dose-dependently results in increased cue-reactivity (CR) responses to alcohol cues in terms of urge to drink [as measured by the Alcohol Visual Analogue Scale (A-VAS)].
  The A-VAS was rated on 11-point anchored Likert-type scales, where 0 is the minimum score (no craving) and 11 is the maximum score (highest craving intensity). The change in the A-VAS score (deltaA-VAS) was used to indicate decrease (-d) or increase (+d) in craving intensity.
Time Frame: approximately 30 minutes after drug administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ghrelin (1 Microg/kg) | Ghrelin (3 Microg/kg) | Saline Solution
Number analyzed (Participants) | 13 | 14 | 18
units on a scale | 1.95 (2.19) | 2.66 (2.19) | 4.29 (2.17)

2. Primary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability.
Description: Whether ghrelin intravenous (i.v.), as compared to saline i.v., does not significantly increase Adverse Events (AEs).
Time Frame: participants will be followed after the cue-reactivity experiment, an expected average of 7 days
Measure: Number; unit: participants
Arm/Group | Ghrelin (1 Microg/kg) | Ghrelin (3 Microg/kg) | Saline Solution
Number analyzed (Participants) | 13 | 14 | 18
participants | 11 | 12 | 15

3. Primary Outcome: Salivation
Description: Whether ghrelin intravenous (i.v.), as compared to saline i.v., dose-dependently results in increased cue-reactivity (CR) responses to alcohol cues in terms of psychophysiological responses, namely salivation changes.
Time Frame: approximately 30 minutes after drug administration
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Ghrelin (1 Microg/kg) | Ghrelin (3 Microg/kg) | Saline Solution
Number analyzed (Participants) | 13 | 14 | 18
gram | 1.8 (1.4) | 1.9 (1.4) | 3.2 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected +17 minutes and +29 minutes after the ghrelin/placebo administration was ended.
Description: The Systematic Assessment for Treatment Emergent Events (SAFTEE) was used for adverse events. For references, see: Levine J, Schooler NR (1986). Psychopharmacology bulletin. 22:343-381; and Johnson BA, Ait-Daoud N, Roache JD (2005). Journal of Studies on Alcohol Supplement.157-167; discussion 140.
Arm/Group | Ghrelin (1 Microg/kg) | Ghrelin (3 Microg/kg) | Saline Solution
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 11/13 | 12/14 | 15/18
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ghrelin (1 Microg/kg) (N=13) | Ghrelin (3 Microg/kg) (N=14) | Saline Solution (N=18)
Increase in appetite (Nervous system disorders) | 8 | 11 | 8
Decrease in appetite (Nervous system disorders) | 0 | 4 | 7
Dizziness (Nervous system disorders) | 0 | 4 | 3
Changes in Vision (Eye disorders) | 0 | 2 | 2
Sleepness (Nervous system disorders) | 2 | 2 | 4
Fatigue (Nervous system disorders) | 2 | 0 | 2
Difficulty with coordination (Nervous system disorders) | 1 | 4 | 3
Difficulty with Concentration (Nervous system disorders) | 0 | 0 | 1
Tingling in Fingers or Toes (Nervous system disorders) | 1 | 0 | 2
Word finding Difficulties (Nervous system disorders) | 0 | 0 | 2
Memory Difficulties (Nervous system disorders) | 0 | 0 | 3
Change in Taste (Nervous system disorders) | 1 | 1 | 2
Tremor (Nervous system disorders) | 1 | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2
Restlessness (Nervous system disorders) | 2 | 1 | 7
Anxiety (Psychiatric disorders) | 7 | 2 | 4
Irritability (Nervous system disorders) | 1 | 1 | 2
Mood Disturbance (Psychiatric disorders) | 0 | 3 | 5
Confusion (Nervous system disorders) | 0 | 1 | 2
Changes in Libido (Reproductive system and breast disorders) | 0 | 0 | 3
Slowed Breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Swelling of throat or tongue (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Difficulty passing urine (Renal and urinary disorders) | 0 | 0 | 1
fast heart beat (Cardiac disorders) | 0 | 0 | 1
Muscle aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
eye pain (Eye disorders) | 0 | 0 | 2
Decreased sweating (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Small proof-of-concept study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No